CLINICAL TRIAL: NCT03611270
Title: Clinical Evaluation of the Therapeutic Intra-Vascular Ultrasound (TIVUS™) System for Pulmonary Artery Denervation in Patients With Pulmonary Hypertension Due to Left Heart Disease
Brief Title: TReatment of Pulmonary Hypertension Group II Study
Acronym: TROPHY-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SoniVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNS02-001
Record Dates: First submitted 2018-06-20; First posted 2018-08-02 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Hypertension (PH) Due to Left Heart Disease
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Pulmonary Denervation — Pulmonary Denervation (PDN) using the TIVUS™ System will be performed in patient suffering from pulmonary hypertension after completion of screening and eligibility phase, The procedure will be performed during right heart catheterisation. Safety and effectiveness of the PDN treatment will be assessed during one year follow up.

SUMMARY:
The objective of this study is to assess the safety and initial effectiveness of the TIVUS™ System when used for pulmonary artery denervation in group II PH patients through change in clinical parameters including hemodynamics, exercise tolerance, and quality of life.

This is a prospective, multi-center, non-randomized, open-label clinical trail. The study will be conducted in up to 3 centers and will recruit up to 15 patients diagnosed with pulmonary hypertension due to left heart disease that demonstrate combined pre and post capillary involvement with PVR>3 wood units.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study obtained from the patient, according to local regulations, prior to initiation of any study mandated procedure.
* Male or female, ≥ 18 years of age at the time of screening
* Patient with known pulmonary hypertension (PH) due to left heart disease (WHO Group II) diagnosed as either HFpEF or HFrEF at chronic state receiving stable guideline directed medical therapy.
* Combined post-capillary and precapillary pulmonary hypertension diagnosis confirmed by hemodynamic evaluation performed prior to screening or during baseline (Eligibility II visit) procedure
* Patient with a current diagnosis of NYHA functional class II/III
* Patient with eGFR levels of ≥ 30 ml/min/1.73m2or serum creatinine levels of ˂ 150μmol/l

Exclusion Criteria:

* Pregnant women or women planning a pregnancy within 12 months of study enrolment
* Patient with significant co-morbid condition(s) which, at the discretion of the PI, are deemed to prohibit study entry
* Patient with life expectancy of less than a year
* Concurrent enrollment in another device or drug trial except for observational studies (unless specifically approved by the sponsor)
* Patient with pulmonary artery anatomy that precludes treatment
* Patient with moderate to severe pulmonary artery stenosis
* Patient with any pulmonary artery aneurysm
* Patient who has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident in the previous 6 months
* Patient experiencing a current episode of acute decompensated heart failure
* Patient who has cardiac pacemakers/ICD/CRT-D that were implanted fewer than three months prior to enrolment. Patient who has implantable Cardiomems device, neurostimulators or drug infusion devices, regardless of implant date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Procedural related Adverse Events (complications) at up to 30 days post procedure | 30 days
  Procedural related Adverse Events (complications) at up to 30 days post procedure including pulmonary artery perforation/dissection, acute thrombus formation in the pulmonary artery, pulmonary artery aneurysm, vascular stenosis, hemoptysis, all cause PH related as well as procedural related death.

SECONDARY OUTCOMES:
Changes in cardiopulmonary exercise test | 4 month
  Changes in cardiopulmonary exercise test (CPET) results (Peak VO2, VE/VCO2 slope, VO2 at anaerobic threshold, peak workload) from baseline
Change in resting mean right atrial pressure | 4 month
  Change in resting mean atrial pressure (mRAP) from baseline
Changes in 6MWD from baseline | 4 month
  Changes in 6MWD from baseline
Changes in Echocardiography parameters | 4 month
  Changes in Echocardiography parameters including Right Ventricular function from baseline
Change in NT-BNP levels | 4 month
  Change in NT-BNP levels from baseline
Procedure related and PH worsening adverse events | 12 month
  Procedure related and PH worsening adverse events and all cause death up to 12 months will be recorded, and serious adverse events will be reported in accordance with regulatory requirements.
Change in exercise mean right atrial pressure | 4 month
  Change in exercise mean right atrial pressure (mRAP) from baseline
Change in exercise mean pulmonary artery pressure | 4 month
  Change in exercise mean pulmonary artery pressure (mPAP) from baseline
Change in exercise pulmonary vascular resistance | 4 month
  Change in exercise pulmonary vascular resistance (PVR) from baseline
Change in exercise cardiac index | 4 month
  Change in exercise cardiac index (CI) from baseline
Change in resting mean pulmonary artery pressure | 4 month
  Change in resting mean pulmonary artery pressure (mPAP) from baseline
Change in resting pulmonary vascular resistance | 4 month
  Change in resting pulmonary vascular resistance (PVR) from baseline
Change in resting cardiac index | 4 month
  Change in resting cardiac index (CI) from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC San Diego Medical Center, San Diego, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided